CLINICAL TRIAL: NCT01558973
Title: Functional Magnetic Resonance Imaging of Stress and Addictive Disorders
Brief Title: FMRI of Stress and Addictive Disorders
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Other Study IDs: 0405026787; 2P50DA016556-08 (NIH)
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine Dependence; Opioid Dependence; Alcoholism; Pathological Gamblers; Adolescents
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Cocaine dependent
- Opioid dependent
- Alcohol dependent
- Healthy controls
- Adolescents
- Pathological gamblers

SUMMARY:
The purpose of this study is to explore whether frontal brain activation in response to stress varies as a function of the presence or extent of early trauma and whether or not this effect is greater in women compared to men. To examine the effect of stress on thinking and remembering. To examine the separate and interactive effects of stress, addiction, withdrawal, and genetics; and to examine fMRI brain activation associated with stressful, reward-related-cue and neutral/relaxing audiotaped scripts,visual images and emotional video clips in addicted individuals and in healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 13-50 years old (adolescents 13-17 years old)
* Able to read and write.
* COCAINE DEPENDENT SUBJECTS: meet DSM-IV criteria for cocaine dependence; report current cocaine use of at least once a week or more; confirmation of cocaine use via positive urine toxicology screen during initial assessments and upon admission to the CNRU.
* OPIOID DEPENDENT SUBJECTS: meet DSM-IV criteria for opiate dependence and are participating in substance abuse treatment including pharmacotherapy for opioid dependence.
* ALCOHOL DEPENDENT SUBJECTS: meet DSM-IV criteria for alcohol dependence and are currently abstinent from alcohol as documented by substance abuse treatment participation.
* HEALTHY CONTROLS: negative urine toxicology screens during intake appointments indicating no history of current or past dependence on alcohol or illicit drug use.
* Healthy adolescent boys and girls, with no medical or psychiatric conditions;
* WOMEN: have a regular menstrual cycle.

Exclusion Criteria:

* CONTROLS: lifetime or current history of any substance abuse/dependence (excluding nicotine).
* Regular use of any psychoactive drugs including anxiolytics and antidepressants.
* Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, liver, thyroid pathology; subjects on medications for any medical condition will be excluded.
* Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded including subjects who work as welders.
* Women on oral contraceptives, peri- and post-menopausal women, and pregnant or lactating women (as alterations in stress response are associated with these states).
* IQ below 75

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cocaine dependent individuals, opioid dependent individuals, alcohol dependent individuals, healthy controls, adolescent subjects, pathological gamblers
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2005-08; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Neural responses to change will be measured. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States